CLINICAL TRIAL: NCT06224283
Title: Confronto Tra Radiomica e i Criteri Convenzionali di Risposta Nella Previsione Della Progressione Del Tumore Desmoide Dopo Crioablazione
Brief Title: Radiomics Compared With Conventional Response Criteria for Predicting Progression of Desmoid Tumor After Cryoablation
Acronym: Cryomics
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor
Other Study IDs: CE AVEC: 570/2023/Oss/IOR
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Desmoid
MeSH Terms: conditions — Desmoid Tumors | interventions — Cryosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Performed cryotherapy: Patients who received cryoablation for desmoid tumor and no chemotherapy
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Cryoablation — Cryoablation, a technique used in interventional radiology, involves repeated cycles of freezing, leading to cell death. Recent studies showed that percutaneous image-guided cryoablation appears to be safe and effective for local control for patients with extra-abdominal desmoid tumors

SUMMARY:
Desmoid tumors (DT) are uncommon tumors that arise from musculoaponeurotic structures. Despite benign, they can cause pain and disability due to their tendency to be locally aggressive. Cryoablation, a technique used in interventional radiology, has gained popularity in recent years as a treatment option for sporadic DT. This involves repeated cycles of freezing, leading to cell death. Recent studies showed that percutaneous image-guided cryoablation appears to be safe and effective for local control for patients with extra-abdominal desmoid tumors.Although changes in the heterogeneity of tumors are commonly known, they are often ignored in response criteria that only evaluate tumor size in a single dimension, such as Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Nevertheless, MRI can reveal early changes in tumor heterogeneity in responding tumors, resulting from a reduction in cellular area and an increase in fibro-necrotic content, before any dimensional changes occur. These changes in heterogeneity can be quantified using a radiomics approach. The aim of this study is to develop radiomics response criteria dedicated to the evaluation of DT treated with cryoablation as a first line treatment and to compare their performance with those of alternative radiologic response criteria for predicting progression according to RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

* desmoid tumor treated at Rizzoli Orthopaedic Institute with cryoablation
* baseline MRI
* clinical and radiologic follow-up until disease progression or the start of a new line of treatment performed every 3 months, with a minimum of 6 months follow-up

Exclusion Criteria:

- not meeting inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were treated with cryoablation for desmoid tumor
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression of disease using mRECIST 1.1 criteria | 6 months
  The aim of this study is to develop radiomics response criteria dedicated to the evaluation of DT treated with cryoablation based on quantification of early changes in heterogeneity sign at MRI images and to compare their performance with those of alternative radiologic response criteria for predicting progression according to mRECIST 1.1.
  Description of mRECIST 1.1 criteria: CR = complete response, disappearing of contrast enhancement of all lesions; PR= partial response, ≥30% dicrease in the sum of the diameters of contrast enhancement of target lesions; SD= stable disease, neither partial response nor progressive disease; PD= progressive disease, ≥20% size increase in contrast enhancement of the target lesions or new disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Giancarlo Facchini, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auloge P, Garnon J, Robinson JM, Thenint MA, Koch G, Caudrelier J, Weiss J, Cazzato RL, Kurtz JE, Gangi A. Percutaneous cryoablation for advanced and refractory extra-abdominal desmoid tumors. Int J Clin Oncol. 2021 Jun;26(6):1147-1158. doi: 10.1007/s10147-021-01887-y. Epub 2021 Mar 11. PMID 33709291
- [Background] Limkin EJ, Sun R, Dercle L, Zacharaki EI, Robert C, Reuze S, Schernberg A, Paragios N, Deutsch E, Ferte C. Promises and challenges for the implementation of computational medical imaging (radiomics) in oncology. Ann Oncol. 2017 Jun 1;28(6):1191-1206. doi: 10.1093/annonc/mdx034. PMID 28168275